CLINICAL TRIAL: NCT01714466
Title: Pharmacodynamic and Clinical Evaluation of Dose and Taste-optimised Low Volume PEG-based Bowel Cleansing Solutions Using the Split-dosing Intake Regimen in Healthy Subjects and in Subjects Undergoing Screening Colonoscopy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Norgine (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NER1006-01/2012 (OPT)
Record Dates: First submitted 2012-10-19; First posted 2012-10-26 (Estimated); Last update posted 2014-11-20 (Estimated); Status verified 2014-11

CONDITIONS: Colon Cancer
MeSH Terms: conditions — Colonic Neoplasms | interventions — MoviPrep

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (8):
- Part A, arm 1 (Experimental): Evening dose of TF048. Morning dose of TF043
  Interventions: Drug: NER1006
- Part A, arm 2 (Experimental): Evening dose of TF043. Morning dose of TF048
  Interventions: Drug: NER1006
- Part A, arm 3 (Experimental): Evening dose of TF047. Morning dose of TF043
  Interventions: Drug: NER1006
- Part A, arm 4 (Active Comparator): MOVIPREP (Both evening and morning dose)
  Interventions: Drug: MOVIPREP
- Part B, arm 1 (Experimental): IMP selected based on the optimal dosing sequence and volume identified from Part A
  Interventions: Drug: NER1006
- Part B, arm 2 (Experimental): IMP as used in Part B, arm 1, with a differing amount of additional clear fluid being consumed
  Interventions: Drug: NER1006
- Part B, arm 3 (Active Comparator): IMP as used in Part B, arm 1, except for a reduced amount of ascorbate
  Interventions: Drug: NER1006
- Part B, arm 4 (Experimental): MOVIPREP used in both evening and morning dose
  Interventions: Drug: MOVIPREP

INTERVENTIONS:
Drug: NER1006
  Arms: Part A, arm 1; Part A, arm 2; Part A, arm 3; Part B, arm 1; Part B, arm 2; Part B, arm 3
Drug: MOVIPREP
  Arms: Part A, arm 4; Part B, arm 4

SUMMARY:
A study to assess the pharmacodynamics, safety and tolerability of a PEG-based bowel cleansing solution (MOVIPREP®)

ELIGIBILITY:
Inclusion Criteria:

* The subject's written informed consent must be obtained prior to inclusion.
* Subjects age 40 to 70 years.
* Part B only: Subjects willing to undergoing a screening colonoscopy, where the subject:

  1. is between 40 and 70 years of age and has a known personal or familial risk of colon neoplasia,or
  2. is aged 55 to 70.
* Part A: Subjects need to be without any history of clinically significant gastrointestinal symptoms by clinical judgement and without the presence of acute abdominal discomfort or symptoms.
* Females of child bearing potential must be surgically sterile, post- menopausal, practicing true sexual abstinence or using an acceptable form of effective contraception throughout the study from the following list: contraceptive injections, implants, oral contraceptives, intrauterine system (IUS), some intrauterine devices (IUDs), vasectomised partner or barrier method (condom or occlusive cap) with spermicidal foam/gel/film/cream/suppository. Females using oral contraceptives must also use additional contraception. Hormonal and IUD methods of contraception must be established for a period of 3 months prior to dosing and cannot be changed or altered during the study. All females must have a negative pregnancy test at screening and check-in (unless post-menopausal).
* Willing, able and competent to complete the entire procedure and to comply with study instructions.
* Ferrous sulphate should be stopped at least one week prior to study medication.

Exclusion Criteria:

* Part A only: Subjects undergoing screening colonoscopy.
* Presence of current clinically significant functional gastrointestinal (GI) disorder (e.g. gastric emptying disorder, chronic constipation, irritable bowel syndrome [IBS]).
* Regular use of laxatives or colon motility altering drugs in the last month.
* Donation or loss of 500 mL or more of blood within 8 weeks prior to the first dose of investigational drug.
* Any history or current presence of ileus, gastrointestinal (GI) obstruction or perforation , GI tract cancer, inflammatory bowel disease (IBD) or colonic resection.
* Known glucose-6-phosphatase dehydrogenase deficiency.
* Known phenylketonuria.
* History or evidence of any clinical significant cardiovascular or neurological disease, cardiac, renal or hepatic insufficiency.
* Known hypersensitivity to polyethylene glycols and/or ascorbic acid.
* History or evidence of any clinically relevant electrocardiogram (ECG) abnormalities and/or uncontrolled hypertension.
* Evidence of dehydration.
* Any evidence for clinically significant abnormal sodium or potassium levels or other clinically significant plasma electrolyte disturbances.
* Females who are not post-menopausal with a positive pregnancy test. Females not using reliable methods of birth control if not post-menopausal.
* Clinically relevant findings on physical examination based on the Investigator's judgement.
* Clinically relevant deviations of laboratory parameters from reference ranges at screening or check-in evaluation.
* Positive serology for chronic viral hepatitis or human immunodeficiency virus (HIV) at screening.
* History of drug or alcohol abuse within the 12 months prior to dosing or evidence of such abuse as indicated by the laboratory assays conducted during the screening or check-in evaluations.
* Subjects who are unwilling to comply with the provisions of the study protocol.
* Concurrent participation in an investigational drug study or participation within 3 months of study entry.
* Subject has a condition or is in a situation, which in the Investigator's opinion may put the subject at significant risk, may confound the study results, or may interfere significantly.
* Previous participation in the study.
* Persons who are ordered to live in an institution on court or authority order

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Actual)
Dates: Start 2012-10; Primary Completion 2013-07 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Stool weight output | 36 hours post-dose
  Stool weight output generated by the IMP from the start of the intake on the evening of Day 1 and the following 24 hours
Cleansing success rate | 36 hours post-dose
  The cleansing success rate (grade A or B according to the Harefield Cleansing Scale)

SECONDARY OUTCOMES:
Tolerability of medication (vomiting rate) | 36 hours post-dose
  The patient's tolerability to the study medication by measuring their vomiting rate for both parts A and B
EQ 5D patient questionnaire outcome (Part A only) | 36 hours post-dose
  Patients to use the EQ 5D patient questionnaire to assess their study medication for part A
Cleansing scores for each colon segment | 36 hours post-dose
  The segmental cleansing scores for each of the five colon segments
Time and volume of IMP to reach a clear effluent | 36 hours post-dose
  The time and volume taken for the IMP to reach a clear effluent
Ascorbate concentration | 36 hours post-dose
  Concentration of ascorbate components and its metabolites (such as dehydroascorbic acid and oxalic acid)
Electrolytes concentration | 36 hours post-dose
  Concentration of electrolytes in blood, urine and faeces
PEG3350 concentration | 36 hours post-dose
  Presence of PEG3350 in faeces, at defined time points, to demonstrate biological activities

CONTACTS AND LOCATIONS:
Overall Officials: Rudiger Kornberger, MD, Principal Investigator — Parexel
Locations (2):
- Germany (2):
  - PAREXEL International Early Product Development Unit, Berlin
  - Parexel International GmbH, Berlin

REFERENCES:
- [Derived] Clayton LB, Tayo B, Halphen M, Kornberger R. Novel 1 L polyethylene glycol-based bowel preparation (NER1006): proof of concept assessment versus standard 2 L polyethylene glycol with ascorbate - a randomized, parallel group, phase 2, colonoscopist-blinded trial. BMC Gastroenterol. 2019 May 30;19(1):79. doi: 10.1186/s12876-019-0988-y. PMID 31146679